CLINICAL TRIAL: NCT00737997
Title: Effect of Early Administration of Morphine on the Development of Acute Opioid Tolerance During Infusion of Remifentanil for Pediatric Scoliosis Surgery
Brief Title: Effect of Early Morphine Administration on the Development of Acute Opioid Tolerance During Pediatric Scoliosis Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Mark Crawford, Anesthesiologist-In-Chief, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000009741
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Scoliosis
Keywords: Pediatrics; Scoliosis; Morphine; Surgery; Analgesia
MeSH Terms: conditions — Scoliosis; Agnosia | interventions — Morphine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Other: Saline
- 2 (Experimental)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — 150 mcg/kg diluted in normal saline to a volume of 10 ml at time of induction of anesthesia
  Arms: 2
Other: Saline — 10 ml saline alone
  Arms: 1

SUMMARY:
The purpose of this study is to examine if morphine administered by bolus before initiating Remifentanil by infusion decreases the incidence of acute post-operative opioid tolerance as demonstrated by decreased post - operative morphine consumption in children undergoing scoliosis surgery.

DETAILED DESCRIPTION:
At our institution, a study has recently demonstrated that intraoperative infusion of remifentanil is associated with development of clinically relevant acute opioid tolerance in adolescents undergoing scoliosis surgery. This results in increased morphine consumption which in turn is associated with increased incidence of side effects such as respiratory depression, nausea and vomiting, pruritus, ileus and urinary retention. All of these side effects can result in increased consumption of rescue medications with the additional potential for increased duration of patient stay. Any measures that can be introduced to decrease the development of acute opioid tolerance in this patient population would have significant impact on patient morbidity, patient comfort and possibly duration of patient stay.

ELIGIBILITY:
Inclusion Criteria:

* Unpremedicated
* ASA physical status 1 or 2
* Aged 11 - 18
* Scheduled to undergo posterior instrumentation for correction of idiopathic scoliosis

Exclusion Criteria:

* Chronic opioid use within three months prior to surgery
* Inability to self-administer morphine using a patient-controlled analgesia (PCA) device
* Elective postoperative ventilation
* Obesity (> 130% ideal body weight)
* Known sensitivity to morphine, remifentanil or any other agent within the standardized protocol
* Failure to obtain written consent or assent

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | Every hour for four hours and then every four hours thereafter for 48 hours

SECONDARY OUTCOMES:
Propofol and remifentanil consumption | 48 hours
Incidences of post-operative nausea, vomiting, pruritus and pyrexia | every hour for four hours and then every four hours thereafter for 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mark Crawford, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] McDonnell C, Zaarour C, Hull R, Thalayasingam P, Pehora C, Ahier J, Crawford MW. Pre-treatment with morphine does not prevent the development of remifentanil-induced hyperalgesia. Can J Anaesth. 2008 Dec;55(12):813-8. doi: 10.1007/BF03034052. PMID 19050084